CLINICAL TRIAL: NCT04485364
Title: Place of Circulating Biomarkers and Respiratory Eicosanoids in the Prognosis of Severe Forms of Covid-19 Pneumonia: BioCovid Study
Brief Title: Place of Circulating Biomarkers and Respiratory Eicosanoids in the Prognosis of Severe Forms of Covid-19 Pneumonia
Acronym: BIOCOVID
Status: Completed | Type: Observational
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Collaborators: Versailles Hospital (Other); Centre Hospitalier Victor Dupouy (Other)
Responsible Party: Sponsor
Other Study IDs: BIOCOVID
Record Dates: First submitted 2020-07-23; First posted 2020-07-24 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-03

CONDITIONS: Coronavirus; Covid19
Keywords: eicosanoids; biomarkers; covid19
MeSH Terms: conditions — Coronavirus Infections; COVID-19

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — During the patient's hospitalization, a blood sample will be taken on a citrate tube in addition to the usual samples during the patient's hospital care. A tracheal aspiration will be systematically performed in order to limit patient congestion and the risk of atelectasis.
  These samples will be destroyed after the study.

SUMMARY:
The research is a prospective, multicentric (Groupe hospitalier Paris Saint-Joseph, Centre Hospitalier de Versailles André Mignot and Centre Hospitalier Victor Dupouy), non-interventional, prospective study. It aims at measuring eicosanoids at different stages of Covid-19 infection.

DETAILED DESCRIPTION:
The reason for the involvement of overweight in the severity of viral respiratory pathologies, particularly during influenza and coronavirus infections, has been the subject of numerous studies which have made it possible to objectify the importance of viral load (at least in mice), particularly in the lower airways and in the alveolar sacs, leading to tissue alteration and alveolar haemorrhage. The mechanisms responsible for alveolar damage during viral pathologies, particularly Coronavirus, are very similar to those observed during acute respiratory distress syndromes in adults. In many situations, endotoxin (or lipopolysaccharide, LPS) plays a major role in the pathophysiology and even the severity of respiratory damage, in particular due to the existence of circulating endotoxin from the causative pathogen (Gram-negative bacteria), but also due to translocation of digestive origin in the context of sepsis (systemic inflammatory response) which is associated with (if not responsible for) respiratory aggression. The importance of this mechanism during pulmonary aggression of viral origin is however unknown. This respiratory attack is associated with a major systemic inflammatory response, reported during the course of Covid-19 infection as corresponding to a "cytokine storm". However, the course of the inflammation is poorly understood and its prognostic nature in the occurrence of a secondarily severe form is not yet better illustrated.

The inflammatory reaction (cytokines, eicosanoids, etc.) is an essential process for the elimination of pathogens by the host, but it must be limited in intensity and duration, otherwise it becomes deleterious for the infected organ. In the case of the lungs, it can induce an acute respiratory distress syndrome (ARDS), which can be severe as in Covid-19 patients with complications. It can be hypothesized that in the early stages of infection, these mediators may play a protective role against Covid-19. Inhibition of these mediators may therefore be deleterious as has been observed in subjects who have taken non-steroidal anti-inflammatory drugs (NSAIDs) that inhibit the production of eicosanoids.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged over 18 years
* French-speaking
* Patient whose Covid-19 respiratory infection was confirmed by laboratory tests, PCR and any other commercial or public health tests
* Patient hospitalized in intensive care unit and under invasive mechanical ventilation for less than three days (early inflammatory phase)
* Adult acute respiratory distress syndrome according to the Berlin definition
* Patient on long-term statin therapy regardless of the rationale for treatment (or without treatment for the control group).

Exclusion Criteria:

* Patient/family or "medical" proxy who refuses the patient's participation in the study
* Patient under guardianship or curatorship
* Patient deprived of liberty
* Patient under the safeguard of justice.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient aged over 18 years old who was positively tested to the Covid 19 infection and has been hospitalized in the Intensive care Unit and under invasive mechanical ventilation for less than 3 days.
Sampling Method: Probability Sample
Enrollment: 97 (Actual)
Dates: Start 2020-04-14 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-06-06 (Actual)

PRIMARY OUTCOMES:
Inflammatory response in the evolution of respiratory diseases | 6 months = the study duration
  The importance of the inflammatory response in the evolution of respiratory disease during the the patients' hospital care based on criteria such as:
  * The search for systemic biomarkers: the previous work led by the Saint Joseph Hospital Group team has highlighted the potential interest of biomarkers of inflammation in the diagnosis of infectious pathology as well as in the eventual prognosis of these patients.
  * and the study of the production of eicosanoids and their presence in the systemic circulation and in the respiratory tree.

SECONDARY OUTCOMES:
Impact of the respiratory disease during mechanical ventilation | 6 months = the study duration
  Evolution of respiratory pathology during mechanical ventilation.

CONTACTS AND LOCATIONS:
Locations (1):
- Groupe Hospitalier Paris Saint-Joseph, Paris, France

REFERENCES:
- [Result] Bradley BT, Bryan A. Emerging respiratory infections: The infectious disease pathology of SARS, MERS, pandemic influenza, and Legionella. Semin Diagn Pathol. 2019 May;36(3):152-159. doi: 10.1053/j.semdp.2019.04.006. Epub 2019 Apr 17. PMID 31054790
- [Result] Yin Y, Wunderink RG. MERS, SARS and other coronaviruses as causes of pneumonia. Respirology. 2018 Feb;23(2):130-137. doi: 10.1111/resp.13196. Epub 2017 Oct 20. PMID 29052924
- [Result] Vijayanand P, Wilkins E, Woodhead M. Severe acute respiratory syndrome (SARS): a review. Clin Med (Lond). 2004 Mar-Apr;4(2):152-60. doi: 10.7861/clinmedicine.4-2-152. PMID 15139736
- [Result] Fehr AR, Channappanavar R, Perlman S. Middle East Respiratory Syndrome: Emergence of a Pathogenic Human Coronavirus. Annu Rev Med. 2017 Jan 14;68:387-399. doi: 10.1146/annurev-med-051215-031152. Epub 2016 Aug 26. PMID 27576010